CLINICAL TRIAL: NCT03248375
Title: The Impact of 90Yttrium (Y90) Radiation Segmentectomy on Hepatocellular Carcinoma and Cirrhosis
Brief Title: Impact of Y90 Radiation Segmentectomy on HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Aaron M Fischman, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 15-0980
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Unresectable Hepatocellular Carcinoma; Radioembolization; Radiation Segmentectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Individuals with the targeted medical condition is given the experimental therapy and then followed over time to observe their response.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Radiation Segmentectomy (Other): Radiation Segmentectomy on Resectable HCC
  Interventions: Radiation: Radiation Segmentectomy

INTERVENTIONS:
Radiation: Radiation Segmentectomy — The administration of radioactivity in a branch of an artery of the liver

SUMMARY:
The aim of this pilot study is to assess the efficacy of radiation segmentectomy with Theraspheres in patients with unresectable hepatocellular carcinoma that would qualify for thermal ablation as per the BCLC guidelines, but are unable to receive thermal ablation due to unfavorable location of target lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years, regardless of race or gender
* Hepatocellular Carcinoma confirmed by histology for non-cirrhotic patients or non-invasive criteria according to AASLD for cirrhotic patients
* Child-Pugh class A or B7 without ascites
* Single tumor nodule ≤ 3 cm with a maximum distance of 5 mm from portal vein, hepatic vein, inferior vena cava, diaphragm, heart, stomach, bowel, liver capsule, gallbladder, bile duct
* No prior locoregional treatment or external beam therapy of current HCC (recurrent HCC after resection may be included)
* No confirmed extrahepatic metastases
* No evidence of macrovascular invasion
* ECOG 0
* Albumin > 3.0 g/dL
* PLT ≥ 40 x103/μL
* WBC ≥ 1.5 x103/μL
* AST/ALT ≤ 5 times the upper limit of normal (U/L)
* Creatinine ≤ 2.0 mg /dL
* No indication for any possible curative treatment after multidisciplinary assessment (surgery, ablation)
* No contraindication to angiography or selective visceral catheterization
* No history of severe allergy or intolerance to contrast agents, narcotics, sedatives.
* Negative serum pregnancy test
* Signed informed consent form

Exclusion Criteria:

* Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Fischman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong JB, McQuillan GM, McHutchison JG, Poynard T. Estimating future hepatitis C morbidity, mortality, and costs in the United States. Am J Public Health. 2000 Oct;90(10):1562-9. doi: 10.2105/ajph.90.10.1562. PMID 11029989
- [Background] Yao FY, Ferrell L, Bass NM, Watson JJ, Bacchetti P, Venook A, Ascher NL, Roberts JP. Liver transplantation for hepatocellular carcinoma: expansion of the tumor size limits does not adversely impact survival. Hepatology. 2001 Jun;33(6):1394-403. doi: 10.1053/jhep.2001.24563. PMID 11391528
- [Background] Llovet JM, Mas X, Aponte JJ, Fuster J, Navasa M, Christensen E, Rodes J, Bruix J. Cost effectiveness of adjuvant therapy for hepatocellular carcinoma during the waiting list for liver transplantation. Gut. 2002 Jan;50(1):123-8. doi: 10.1136/gut.50.1.123. PMID 11772979
- [Background] Llovet JM, Bruix J. Systematic review of randomized trials for unresectable hepatocellular carcinoma: Chemoembolization improves survival. Hepatology. 2003 Feb;37(2):429-42. doi: 10.1053/jhep.2003.50047. PMID 12540794
- [Background] Curley SA, Izzo F, Ellis LM, Nicolas Vauthey J, Vallone P. Radiofrequency ablation of hepatocellular cancer in 110 patients with cirrhosis. Ann Surg. 2000 Sep;232(3):381-91. doi: 10.1097/00000658-200009000-00010. PMID 10973388
- [Background] Cheng JC, Wu JK, Lee PC, Liu HS, Jian JJ, Lin YM, Sung JL, Jan GJ. Biologic susceptibility of hepatocellular carcinoma patients treated with radiotherapy to radiation-induced liver disease. Int J Radiat Oncol Biol Phys. 2004 Dec 1;60(5):1502-9. doi: 10.1016/j.ijrobp.2004.05.048. PMID 15590181
- [Background] Dawson LA, Ten Haken RK. Partial volume tolerance of the liver to radiation. Semin Radiat Oncol. 2005 Oct;15(4):279-83. doi: 10.1016/j.semradonc.2005.04.005. PMID 16183482
- [Background] Gaba RC, Lewandowski RJ, Kulik LM, Riaz A, Ibrahim SM, Mulcahy MF, Ryu RK, Sato KT, Gates V, Abecassis MM, Omary RA, Baker TB, Salem R. Radiation lobectomy: preliminary findings of hepatic volumetric response to lobar yttrium-90 radioembolization. Ann Surg Oncol. 2009 Jun;16(6):1587-96. doi: 10.1245/s10434-009-0454-0. Epub 2009 Apr 9. PMID 19357924
- [Background] Young JY, Rhee TK, Atassi B, Gates VL, Kulik L, Mulcahy MF, Larson AC, Ryu RK, Sato KT, Lewandowski RJ, Omary RA, Salem R. Radiation dose limits and liver toxicities resulting from multiple yttrium-90 radioembolization treatments for hepatocellular carcinoma. J Vasc Interv Radiol. 2007 Nov;18(11):1375-82. doi: 10.1016/j.jvir.2007.07.016. PMID 18003987
- [Background] Riaz A, Lewandowski RJ, Kulik LM, Mulcahy MF, Sato KT, Ryu RK, Omary RA, Salem R. Complications following radioembolization with yttrium-90 microspheres: a comprehensive literature review. J Vasc Interv Radiol. 2009 Sep;20(9):1121-30; quiz 1131. doi: 10.1016/j.jvir.2009.05.030. Epub 2009 Jul 29. PMID 19640737
- [Background] Lencioni R, Llovet JM. Modified RECIST (mRECIST) assessment for hepatocellular carcinoma. Semin Liver Dis. 2010 Feb;30(1):52-60. doi: 10.1055/s-0030-1247132. Epub 2010 Feb 19. PMID 20175033
- [Background] Riaz A, Gates VL, Atassi B, Lewandowski RJ, Mulcahy MF, Ryu RK, Sato KT, Baker T, Kulik L, Gupta R, Abecassis M, Benson AB 3rd, Omary R, Millender L, Kennedy A, Salem R. Radiation segmentectomy: a novel approach to increase safety and efficacy of radioembolization. Int J Radiat Oncol Biol Phys. 2011 Jan 1;79(1):163-71. doi: 10.1016/j.ijrobp.2009.10.062. Epub 2010 Apr 24. PMID 20421150
- [Background] Bargellini I, Bozzi E, Campani D, Carrai P, De Simone P, Pollina L, Cioni R, Filipponi F, Bartolozzi C. Modified RECIST to assess tumor response after transarterial chemoembolization of hepatocellular carcinoma: CT-pathologic correlation in 178 liver explants. Eur J Radiol. 2013 May;82(5):e212-8. doi: 10.1016/j.ejrad.2012.12.009. Epub 2013 Jan 15. PMID 23332890
- [Background] Komorizono Y, Oketani M, Sako K, Yamasaki N, Shibatou T, Maeda M, Kohara K, Shigenobu S, Ishibashi K, Arima T. Risk factors for local recurrence of small hepatocellular carcinoma tumors after a single session, single application of percutaneous radiofrequency ablation. Cancer. 2003 Mar 1;97(5):1253-62. doi: 10.1002/cncr.11168. PMID 12599233
- [Background] Golfieri R, Renzulli M, Mosconi C, Forlani L, Giampalma E, Piscaglia F, Trevisani F, Bolondi L; Bologna Liver Oncology Group (BLOG). Hepatocellular carcinoma responding to superselective transarterial chemoembolization: an issue of nodule dimension? J Vasc Interv Radiol. 2013 Apr;24(4):509-17. doi: 10.1016/j.jvir.2012.12.013. Epub 2013 Feb 18. PMID 23428355
- [Derived] Kim E, Sher A, Abboud G, Schwartz M, Facciuto M, Tabrizian P, Knesaurek K, Fischman A, Patel R, Nowakowski S, Llovet J, Taouli B, Lookstein R. Radiation segmentectomy for curative intent of unresectable very early to early stage hepatocellular carcinoma (RASER): a single-centre, single-arm study. Lancet Gastroenterol Hepatol. 2022 Sep;7(9):843-850. doi: 10.1016/S2468-1253(22)00091-7. Epub 2022 May 23. PMID 35617978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were enrolled between Aug 3, 2016, and April 4, 2019
Groups:
- Radiation Segmentectomy: Patients diagnosed with hepatocellular carcinoma underwent radiation segmentectomy on resectable hepatocellular carcinoma and cirrhosis HCC.
  Radiation segmentectomy was done with ⁹⁰Y microspheres infused through selective branches off the hepatic artery. The delivery device used was glass-based (TheraSphere; Boston Scientific, Ottawa, ON, Canada), in which ⁹⁰Y is an integral constituent of the biocompatible glass matrix. Estimated dose to the treated area was >205Gy.
Period: Overall Study
Arm/Group | Radiation Segmentectomy
Started | 29
Completed | 24
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Groups:
- Radiation Segmentectomy: Radiation Segmentectomy on Resectable HCC on patients diagnosed with hepatocellular carcinoma
Arm/Group | Radiation Segmentectomy
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Cause of liver disease [Count of Participants; unit: Participants] — there could be more than one reported cause of liver disease for each participant
  Participants
    Hepatitis B virus | 3
    Hepatitis C virus | 13
    Non-alcoholic steatohepatitis | 5
    Alcohol | 7
    Sarcoidosis | 1
    Haemochromatosis | 1
Child-Pugh score [Count of Participants; unit: Participants] — Total score from 5-15, categorized into Child-Pugh grades A (5 to 6 points), B (7 to 9 points), or C (10 to 15 points). Higher score indicates poorer health outcomes.
  Participants
    A5 | 14
    A6 | 12
    B7 | 3
α-Fetoprotein [Median (Full Range); unit: ng/mL] — Alpha fetoprotein (AFP) is a protein produced by the liver and yolk sac of a developing baby during pregnancy. The normal values in males or nonpregnant females is generally less than 40 micrograms/liter.
  ng/mL | 5 [0 to 409.5]
Albumin-bilirubin grade (ALBI) [Count of Participants; unit: Participants] — ALBI score =0.66×log10 [total bilirubin (µmol/L)] - 0.085× [albumin (g/L)].
  grade 1 (score ≤-2.60)
  grade 2 (-2.60< score ≤-1.39)
  and grade 3 (score >-1.39)
  Lower grade represents better health outcomes.
  Participants
    Albumin-bilirubin grade 1 | 7
    Albumin-bilirubin grade 2 | 22
Ascites [Count of Participants; unit: Participants] | 1
Tumor diameter [Mean (Standard Deviation); unit: cm] | 2.1 (0.4)
Liver segment tumor distribution [Count of Participants; unit: Participants] — Measure refers to the liver segments (1-8 based on Couinaud classification) of tumor location based on pre-treatment imaging
  Participants
    1 - caudate lobe | 0
    2 - left of the left hepatic vein and falciform ligament and superior to the portal plane | 5
    3 - left of the left hepatic vein and falciform ligament and inferior to the portal plane | 0
    4 - between the left and middle hepatic veins - subcardiac location | 8
    5 - located below the portal plane between the middle and right hepatic veins | 2
    6 - located below the portal plane to the right of the right hepatic vein | 5
    7 - located above the portal plane to the right of the right hepatic vein | 3
    8 - located above the portal plane between the middle and right hepatic veins | 11
Location [Count of Participants; unit: Participants] — Central or peripheral location of tumors determined based on pretreatment imaging
  Participants
    Peripheral | 28
    Central | 1
Number of injection locations [Count of Participants; unit: Participants]
  1 | 24
  2 | 5
Lobar volume [Median (Full Range); unit: mL]
  Right | 896.7 [406.7 to 1523.8]
  Left | 439.0 [316.6 to 832.0]
Perfused liver volume [Mean (Standard Deviation); unit: mL] | 153.6 (99.2)
Distribution of Perfused Liver Volumes [Count of Participants; unit: Participants] — Number of patients with perfused liver volumes <100cc, 100-200 cc, and >200cc measured using cone beam CT (CBCT)
  Participants
    <100 cc | 9
    100-200 cc | 12
    >200 cc | 8
Lung shunt fraction (LSF) [Mean (Full Range); unit: percentage reaching lung] — The lung shunt fraction is calculated using macroaggregated albumin (MAA) and performing a nuclear medicine study. It represents the percentage determined by the ratio of the counts in the lungs to the summed counts in the lungs and liver.
  percentage reaching lung | 4 [1.9 to 10.7]
Calculated dose to the perfused segment [Median (Full Range); unit: Gy] — The calculated dose was calculated as a segmental delivery with the goal of more than 205 Gy to the perfused area using the Committee on Medical Internal Radiation Dose model based on tumour response and survival data.
  Gy | 584 [181.0 to 3340.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local Tumor Response According to mRECIST
Description: Efficacy of 90Yttrium (Y90) Radiation Segmentectomy on Unresectable Hepatocellular Carcinoma as measured by tumor response according to mRECIST.
  CR = Disappearance of any intratumoral arterial enhancement in all target lesions PR = At least a 30% decrease in the diameter of the viable (enhancement in the arterial phase) target lesion SD = Any cases that do not qualify for either partial response or progressive disease PD = An increase of at least 20% in the diameter of viable (enhancing) target lesion
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Segmentectomy
Number analyzed (Participants) | 29
Participants
  CR - Complete response | 26
  PR - Partial response | 0
  SD - Stable disease | 0
  PD - Progressive disease | 3

2. Secondary Outcome: Median Time to Progression (TTP)
Description: Time until progression of the target lesion and overall disease based on mRECIST
Time Frame: 2 years
Population: Data for participants who had target lesion progression only
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Radiation Segmentectomy
Number analyzed (Participants) | 3
days | NA [NA to NA] — There was an insufficient number of participants with events to calculate a median TTP. Three patients had target lesion progression at 227, 496, and 668 days.

3. Secondary Outcome: Cumulative Incidence of Participants With Local Progression
Description: Cumulative incidence function estimation of the incidence of the occurrence of local progression (event) at 1 year and 2 years while taking the competing risk of transplant into account.
  Local progression was defined per modified Response Evaluation Criteria In Solid Tumors Criteria (mRECIST) for target lesions and assessed by MRI with local progression defined as an >20% increase in the diameter of the viable (enhancing) target lesion, taking as a reference of the baseline enhancing tumor size.
Time Frame: 1 year and 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation Segmentectomy
Number analyzed (Participants) | 29
percentage of participants
  1 years | 4 [0 to 16]
  2 years | 12 [3 to 28]

4. Secondary Outcome: Quantifying Dose to Target Lesion
Description: The dose was calculated using PET/CT calculated dose estimation delivered to the tumor. Counts on PET/CT post-treatment were used to estimate the dose delivered to the tumor.
Time Frame: 0 days
Population: Dose delivered to the tumour was calculated for 26 (90%) patients with 90Y PET CT imaging. Three (7%) patients were excluded due to technical issues.
Measure: Median (95% Confidence Interval); unit: Gy
Arm/Group | Radiation Segmentectomy
Number analyzed (Participants) | 26
Gy | 1004.6 [844.7 to 1400.8]

5. Secondary Outcome: Number of Treatment-related Adverse Events
Description: Number of treatment related adverse events according to the National Cancer Institute Common Terminology Criteria for Adverse Events v 5.0 (CTCAE).
Time Frame: For 2 years with visits 6 weeks post treatment then every 3 months since treatment for 24 months for assessment of laboratory and clinical symptoms
Measure: Number; unit: events
Arm/Group | Radiation Segmentectomy
Number analyzed (Participants) | 29
events
  fatigue | 9
  nausea, vomiting, or anorexia | 7
  abdominal discomfort | 6
  ascites | 1
  laboratory changes | 24

6. Secondary Outcome: Number of Participants With Access Site-related Adverse Events
Description: Number of participants with access site-related adverse events
Time Frame: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Segmentectomy
Number analyzed (Participants) | 29
Participants
  Arterial injury | 1
  Hematoma (minor) | 4
  None | 24

7. Secondary Outcome: Number of Participants With Treatment-related Laboratory Adverse Events
Description: Number of participants with treatment-related laboratory adverse events assessed 6 weeks post-treatment then every 3 months since treatment for 24 months
Time Frame: For 2 years with visits 6 weeks post treatment then every 3 months since treatment for 24 months for assessment of laboratory changes
Population: All Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Segmentectomy
Number analyzed (Participants) | 29
Participants
  Leukopenia | 13
  Anemia | 3
  Thrombocytopenia | 6
  AST or ALT increased | 4
  ALP increased | 4
  Total blood bilirubin increased | 4
  Albumin decreased | 6
  Creatinine increased | 3
  International normalised ratio increased | 1

ADVERSE EVENTS:
Time Frame: up to 2 years and every 3 months since treatment for 24 months for laboratory changes
Arm/Group | Radiation Segmentectomy
All-Cause Mortality (participants affected / at risk) | 1/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 26/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Segmentectomy (N=29)
Arterial Injury (Injury, poisoning and procedural complications) | 1
Haemotoma (Injury, poisoning and procedural complications) | 4
Fatigue (General disorders) | 9 — Treatment-related
Nausea, Vomiting, or Anorexia (Gastrointestinal disorders) | 7 — Treatment-related
Abdominal discomfort (Gastrointestinal disorders) | 6 — Treatment-related
Ascites (Gastrointestinal disorders) | 1 — Treatment-related
Leukopenia (Blood and lymphatic system disorders) | 13 — Treatment-related laboratory adverse events
Thrombocytopenia (Blood and lymphatic system disorders) | 6 — Treatment-related laboratory adverse events
Anaemia (Blood and lymphatic system disorders) | 3 — Treatment-related laboratory adverse events
AST or ALT increased (Hepatobiliary disorders) | 4 — Treatment-related laboratory adverse events
ALP increased (Hepatobiliary disorders) | 4 — Treatment-related laboratory adverse events
Total blood bilirubin increased (Hepatobiliary disorders) | 4 — Treatment-related laboratory adverse events
Albumin decreased (Metabolism and nutrition disorders) | 6 — Treatment-related laboratory adverse events
Creatinine increased (Investigations) | 3 — Treatment-related laboratory adverse events
International normalised ratio increased (Investigations) | 1 — Treatment-related laboratory adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT03248375/Prot_SAP_000.pdf